CLINICAL TRIAL: NCT02208570
Title: Predictability of the Pulse Pressure Variation During Spontaneous Ventilation on the Incidence of Hypotension During Induction of Anesthesia
Brief Title: Predictability of the Pulse Pressure Variation (PPV) During Spontaneous Ventilation on the Incidence of Hypotension During Induction of Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Hyon Bahk, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JHBahk_PPV_predictability
Record Dates: First submitted 2014-07-14; First posted 2014-08-05 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Hypotension
Keywords: Hypotension during anesthesia induction
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (4):
- P(+)V(+) (Experimental): PPV>14% before anesthesia induction, HES 6ml/kg infused
  Interventions: Other: PPV>14%; Drug: Volume loading
- P(+)V(-) (Experimental): PPV>14% before anesthesia induction, no additional volume infused
  Interventions: Other: PPV>14%
- P(-)V(+) (Experimental): PPV<14% before anesthesia induction, HES 6ml/kg infused
  Interventions: Drug: Volume loading; Other: PPV<14%
- P(-)V(-) (Experimental): PPV<14% before anesthesia induction, no additional volume infused
  Interventions: Other: PPV<14%

INTERVENTIONS:
Other: PPV>14% — Patients whose preoperative pulse pressure variation during spontaneous ventilation exceed 14
  Arms: P(+)V(+); P(+)V(-)
Drug: Volume loading — Hydroxyethyl starch solution 6ml/kg iv injection
  Arms: P(+)V(+); P(-)V(+)
Other: PPV<14% — Patients whose preoperative pulse pressure variation during spontaneous ventilation does not exceed 14
  Arms: P(-)V(+); P(-)V(-)

SUMMARY:
The purpose of this study is to find out the predictability of the pulse pressure variation during spontaneous ventilation on the incidence of hypotension during induction of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing general anesthesia induction with intravenous anesthesia using propofol and remifentanil
* Patients requiring invasive arterial blood pressure monitoring for the surgery

Exclusion Criteria:

* Refusal of consent
* Patients with heart disease (symptomatic valvular heart disease, intracardiac shunt, pulmonary hypertension with pulmonary systolic arterial pressure exceeding 40mmHg)
* FEV1 ≤ 50% predicted FEV1
* Patients with chronic renal failure
* ASA class IV, V, VI
* Systolic arterial blood pressure below 90mmHg before induction of anesthesia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Changes of heart rate and systolic arterial blood pressure from baseline values immediately before tracheal intubation | Three minutes after anesthesia agent injection
  First, we measure the baseline heart rate and systolic arterial blood pressure and calculate the baseline heart rate and blood pressure.
  At 3 minutes after anesthesia agent injection we record the heart rate and blood pressure, and perform endotracheal intubation. Then we calculate the percentile change of blood pressure and heart rate from the baseline values.

SECONDARY OUTCOMES:
Changes of heart rate and systolic arterial blood pressure from baseline values, three minutes before intubation | Three minutes before endotracheal intubation
  We collect the patient's vital signs for 1 second interval during anesthesia induction. We collect the patient's heart rate and blood pressure values for three minutes before endotracheal intubation, and average the numbers. Then we compare the numbers from the baseline value and calculate the changes.
Changes of heart rate and systolic arterial blood pressure from baseline values, three minutes after intubation | Three minutes after endotracheal intubation
  We collect the patient's vital signs for 1 second interval during anesthesia induction. We collect the patient's heart rate and blood pressure values for three minutes after endotracheal intubation, and average the numbers. Then we compare the numbers from the baseline value and calculate the changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea